CLINICAL TRIAL: NCT02621489
Title: Effects on Re-endothelialisation With Bydureon Treatment Add on to Insulin Versus Insulin Alone, Both in Combination With Metformin in Type 2 Diabetic Subjects
Brief Title: Effects on Re-endothelialisation With Bydureon Treatment in Type 2 Diabetes Subjects
Acronym: Rebuild
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Thomas Nystrom, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BY2015
Record Dates: First submitted 2015-11-22; First posted 2015-12-03 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Atherosclerosis; Diabetes; Restenosis
Keywords: Glucagon-like peptide-1; Endothelialization; Cardiac Function; Exenatide; Optical Coherence Tomography
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus | interventions — Exenatide; Insulin Aspart; Metformin; Biguanides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bydureon 2 mg Once Weekly (Experimental): Patients randomised to Bydureon will be treated with Metformin 1g BID, and only receive 10U of Humulin kwickpen QD at bedtime, with no more up-titration of insulin during the study.
  Interventions: Drug: Bydureon; Drug: Humulin kwickpen; Drug: Metformin
- Humulin kwickpen (Active Comparator): Patients randomised to the comparator group will be treated with Meformin 1g BID and Humulin kwickpen to reach a fP-glucose level of 6 mmol/l. For that reason patients will be instructed to increase the bedtime Insulin dose of 2-4U every third day until this goal is reached.
  Interventions: Drug: Humulin kwickpen; Drug: Metformin

INTERVENTIONS:
Drug: Bydureon — 2 mg Once Weekly
  Other Names: Exenatide
  Arms: Bydureon 2 mg Once Weekly
Drug: Humulin kwickpen — Humulin kwickpen 10U QD at bedtime
  Other Names: Insulin Aspart
Drug: Metformin — Metformin 1g BID
  Other Names: Biguanide

SUMMARY:
The aim of the study is to use Exenatide long-acting release (LAR) [Bydureon] to minimize vascular remodeling and neointima formation after Percutaneous Coronary Intervention (PCI) and to accelerate stent endothelialisation.

DETAILED DESCRIPTION:
Exenatide LAR will be given as a once-weekly (s.c.) dose of Bydureon (2 mg) add on to Insulin in combination with Metformin. If patients are Insulin naïve (both groups) an initial dose of 10U (s.c.) at bedtime will be started, and further up-titrated to achieve a fP-glucose levels at 6 mmol/l. Standard care for post myocardial infarction will be given after PCI.

Primary objectives:

To test whether Bydureon, add on to Insulin Neutral Protamine Hagedorn (NPH) + Metformin, is superior vs. Insulin NPH + Metformin alone, in covered stent struts

Secondary objectives:

To test whether Bydureon, add on to Insulin NPH + Metformin, is superior vs. Insulin NPH + Metformin alone: in cardiac and endothelial functions

ELIGIBILITY:
Inclusion Criteria:

1. Patients eligible for PCI with application of DES, due to ACS.
2. Patients with known or newly diagnosed T2D (type 2 diabetes is diagnosed according to current WHO criteria or by the use of anti-diabetic drugs)
3. Male and female subjects 18-80 years.
4. HbA1c (accordingly to IFCC) 47 mmol/mol - 110 mmol/mol.
5. Signed informed consent form.

Exclusion Criteria:

1. Type 1 diabetes (autoantibody positive).
2. Any history of receiving GLP-1 analogues or dipeptidyl peptidase inhibitors within 6 months
3. Known severe heart failure, classified as NYHA 4.
4. Active myocarditis; malfunctioning artificial heart valve.
5. History of ventricular tachycardia within 3 months before study entry; second- or third-degree atrioventricular block.
6. Supine systolic blood pressure <85 mm Hg or >200 mm Hg at screening.
7. Primary renal impairment, creatinine clearance < 45 ml/min if treated with metformin.
8. Uncorrected hypokalemia or hyperkalemia (potassium <3.5 mmol/l or >5.5 mmol/l).
9. Significant anemia (Hb < 90 g/l)
10. Severe gastrointestinal disease, including gastroparesis. As judged by the Investigator.
11. Body mass index (BMI) > 45 kg/m2.
12. Malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy in the previous 5 years. Patients with intraepithelial squamous cell carcinoma of the skin treated with topical 5FU and subjects with basal cell skin cancer are allowed to enter the trial.
13. Females of child bearing potential who are pregnant, breast-feeding or intend to become pregnant.
14. Current drug and alcohol abuse.
15. History of acute or chronic pancreatitis
16. Subjects considered by the Investigator to be unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-12; Primary Completion 2022-08 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
The degree of non-covered stent struts by Bydureon add on to Insulin over that of Insulin as analyzed by optical coherence tomography (OCT). | 12 weeks

SECONDARY OUTCOMES:
Fractional Flow Reserve (FFR) | 12 weeks
  FFR is a unitless index calculated as the ratio between distal coronary and aortic pressure during maximum hyperemia.
Coronary Flow velocity Reserve (CRF) | 12 weeks
  CFR is a unitless index calculated as the ratio between the the mean transit time recorded at maximum hyperemia and at baseline using the thermodilution.
Index of Microcirculatory Resistance (IMR) | 12 weeks
  IMR is a unitless index calculated by dividing the mean distal coronary pressure by the inverse of the mean transit time recorded using the thermodilution technique during maximum hyperemia
Fractional flow reserve positive re-stenosis | 12 weeks
Target lesion failure | 12 weeks
  Need of unplanned PCI in the treated stenosis or significant re-stenosis in the follow-up
Acute coronary syndrome (ACS) and/or repeat revascularization | 12 weeks
Late lumen loss/neointima thickness measured with OCT | 12 weeks
Change in minimal lumen area by OCT | 12 weeks
Left ventricular systolic and diastolic function assessed by echocardiography | 12 weeks
Recovery from endothelial damage, measured by high resolution ultrasound, after PCI | 12 weeks
  Non-invasive ultrasound over the radialis artery after the PCI procedure using Standard 6-7F guiding catheters.
Plasma markers of endothelial activation i.e., E-Selectin, VCAM-1, ICAM-1, nitrotyrosine levels | 12 weeks
Plasma markers of inflammation i.e., CRP, IL-1β, IL-6 and IL-8. | 12 weeks
Plasma markers of matrix remodeling enzymes i.e., MMP-2 and MMP9 | 12 weeks
Circulating endothelial progenitor cells | 12 weeks
Gene expression (Affymetrix) e.g., transcription factors of sirtuins (SIRT) and nitric oxide synthase (NOS) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nyström, Principal Investigator — Karolinska Institutet
Locations (1):
- Dept of clinical science and education Karolinska Institutet Södersjukhuset, Stockholm, Other, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eriksson L, Saxelin R, Rohl S, Roy J, Caidahl K, Nystrom T, Hedin U, Razuvaev A. Glucagon-Like Peptide-1 Receptor Activation Does not Affect Re-Endothelialization but Reduces Intimal Hyperplasia via Direct Effects on Smooth Muscle Cells in a Nondiabetic Model of Arterial Injury. J Vasc Res. 2015;52(1):41-52. doi: 10.1159/000381097. Epub 2015 May 7. PMID 25966620
- [Result] Erdogdu O, Eriksson L, Xu H, Sjoholm A, Zhang Q, Nystrom T. Exendin-4 protects endothelial cells from lipoapoptosis by PKA, PI3K, eNOS, p38 MAPK, and JNK pathways. J Mol Endocrinol. 2013 Mar 18;50(2):229-41. doi: 10.1530/JME-12-0166. Print 2013 Apr. PMID 23343509
- [Result] Erdogdu O, Nathanson D, Sjoholm A, Nystrom T, Zhang Q. Exendin-4 stimulates proliferation of human coronary artery endothelial cells through eNOS-, PKA- and PI3K/Akt-dependent pathways and requires GLP-1 receptor. Mol Cell Endocrinol. 2010 Aug 30;325(1-2):26-35. doi: 10.1016/j.mce.2010.04.022. Epub 2010 May 7. PMID 20452396
- [Result] Erdogdu O, Eriksson L, Nystrom T, Sjoholm A, Zhang Q. Exendin-4 restores glucolipotoxicity-induced gene expression in human coronary artery endothelial cells. Biochem Biophys Res Commun. 2012 Mar 23;419(4):790-5. doi: 10.1016/j.bbrc.2012.02.106. Epub 2012 Feb 27. PMID 22390929
- [Result] Nystrom T, Gutniak MK, Zhang Q, Zhang F, Holst JJ, Ahren B, Sjoholm A. Effects of glucagon-like peptide-1 on endothelial function in type 2 diabetes patients with stable coronary artery disease. Am J Physiol Endocrinol Metab. 2004 Dec;287(6):E1209-15. doi: 10.1152/ajpendo.00237.2004. Epub 2004 Sep 7. PMID 15353407
- [Result] Dokken BB, Piermarini CV, Teachey MK, Gura MT, Dameff CJ, Heller BD, Krate J, Ashgar AM, Querin L, Mitchell JL, Hilwig RW, Kern KB. Glucagon-like peptide-1 preserves coronary microvascular endothelial function after cardiac arrest and resuscitation: potential antioxidant effects. Am J Physiol Heart Circ Physiol. 2013 Feb 15;304(4):H538-46. doi: 10.1152/ajpheart.00282.2012. Epub 2012 Dec 15. PMID 23241323
- [Result] Guagliumi G, Sirbu V, Bezerra H, Biondi-Zoccai G, Fiocca L, Musumeci G, Matiashvili A, Lortkipanidze N, Tahara S, Valsecchi O, Costa M. Strut coverage and vessel wall response to zotarolimus-eluting and bare-metal stents implanted in patients with ST-segment elevation myocardial infarction: the OCTAMI (Optical Coherence Tomography in Acute Myocardial Infarction) Study. JACC Cardiovasc Interv. 2010 Jun;3(6):680-7. doi: 10.1016/j.jcin.2010.04.005. PMID 20630463
- [Derived] Santos-Pardo I, Witt N, Angeras O, Nystrom T. Effects of exenatide on coronary stent's endothelialization in subjects with type 2 diabetes: a randomized controlled trial. The Rebuild study. Cardiovasc Diabetol. 2023 Dec 8;22(1):337. doi: 10.1186/s12933-023-02071-4. PMID 38066597